CLINICAL TRIAL: NCT04254887
Title: EPBD+Small EST VS. Large EST in Patients With Choledocholithiasis Complicated With Duodenal Papillary Diverticula
Brief Title: Effect of EPBD in ERCP on the Prognosis of Patients With Choledocholithiasis Complicated With Duodenal Papillary Diverticula
Acronym: EPBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ERCP-0002
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-10

CONDITIONS: Periampullary Diverticula
Keywords: EPBD

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPBD (Experimental): Small incision of the duodenal nipple + EPBD
  Interventions: Procedure: EPBD
- EST (Active Comparator): Large incision of the duodenal nipple
  Interventions: Procedure: EST

INTERVENTIONS:
Procedure: EPBD — Small incision of the duodenal nipple + EPBD
  Arms: EPBD
Procedure: EST — Large incision of the duodenal nipple + EPBD
  Arms: EST

SUMMARY:
The investigators hypothesized that nipple balloon dilatation could make ERCP more successful and reduce postoperative complications and mortality. So the investigators design this experiment on this assumption.

DETAILED DESCRIPTION:
The incidence of periampullary diverticula in patients with choledocholithiasis is very high at 47.1%. A large number of literatures refered that duodenal papillary diverticulum is a high risk factor for postoperative complications and recurrence of choledocholithiasis . Till now, there have been no randomized controlled trials to explore the effect of nipple balloon dilatation (EPLBD) on the treatment and prognosis of patients with choledocholithiasis complicated with periampullary diverticula (found during ERCP).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with choledocholithiasis. 2. During ERCP, the patient was diagnosed as choledocholithiasis combined with duodenal papillary diverticulum. 3. Ages 16 to 75. 4. choledocholithiasis no larger than 1.5 cm

Exclusion Criteria:

1. Patients with duodenal papillary tumor. 2. Pregnant. 3. Patients with gastrointestinal duct obstruction endoscopy who cannot be operated and who have endoscopic contraindications. 4. Patients with duodenoscopy contraindications. 5. Patients with severe pancreatitis and other serious diseases.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of complications | 1 month
  total complications occurded after operation
time of operation | 1-4 hours
  duration of the ERCP
postoperative recurrent rate | 1 year
  Recurrence rate of choledocholithiasis

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No